CLINICAL TRIAL: NCT07209137
Title: A Single-Group Clinical Trial to Evaluate the Effects of Health Nag's BioActive Collagen Jelly on Skin, Hair, Nail, and Joint Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nag Food Supplement Trading LLC (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20743
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Joint Health; Hair Health; Skin Health
Keywords: Collagen Supplement; Muscle Recovery
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioActive Collagen Jelly Intervention (Experimental): Participants will consume 10 g of BioActive Collagen Jelly daily, on an empty stomach, for 12 weeks.
  Interventions: Dietary Supplement: Dietary Supplement

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — The supplement is intended to support improvements in skin health, hair strength, nail strength, joint health, and overall well-being.

SUMMARY:
This decentralized, single-arm, open-label study evaluates the effects of Health Nag's BioActive Collagen Jelly on skin, hair, nail, and joint health in 40 female participants over 12 weeks. Participants will submit online questionnaires and standardized digital photos, which will be analyzed by dermatology experts.

ELIGIBILITY:
Inclusion Criteria:

* Be female
* Be aged 30-55.
* Anyone who has concerns surrounding their skin health and appearance over the last four weeks.
* Anyone who has concerns surrounding their hair health and hair fall or thinning over the last four weeks.
* Anyone who has been using the same hair and skincare routine and products for at least one month prior to the study, i.e., shampoo, conditioner, products, cleanser, toner, and makeup remover.
* Anyone willing to maintain the same hair and skincare routine and products throughout the 6-month trial, i.e., shampoo, conditioner, products, cleanser, toner, and makeup remover.
* Is willing to discontinue any other supplements or herbal remedies that target skin or hair health including but not limited to collagen.
* Anyone willing to avoid introducing any other supplements, medications, or herbal remedies for the duration of the trial.
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* Resides in the United States.
* Not currently partaking in another research study and will not be partaking in any other research study for the next 6 months and at any point during this study's duration.
* Anyone who owns a smartphone or camera.

Exclusion Criteria:

* Anyone unwilling to follow the study protocol
* Anyone who is planning to undergo facial treatments during the study period, including botox, dermal filler, chemical peels, etc.
* Anyone who has undergone chemical treatments to the hair in the last three months e.g., chemical straightening, hair extensions with chemical bonding, perms, and relaxers.
* Anyone with planned chemical treatments to the hair during the study period, e.g., chemical straightening, hair extensions with chemical bonding, perms, and relaxers.
* Anyone currently taking any prescription medication for hair loss.
* Anyone who has undergone any surgeries or invasive treatments in the last six months or is planning to undergo any surgeries or invasive treatments during the study.
* Anyone who has had any major illness in the last three months.
* Anyone who has any conditions that could affect the hair or scalp (e.g., alopecia areata)
* Anyone who has stopped using hormonal birth control within the past month.
* Anyone who has any chronic skin conditions on the face (e.g., eczema or psoriasis).
* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with any allergies or sensitivities to any of the study product ingredients.
* Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).
* Anyone who is vegan and/or does not consume animal products for any reason.
* Anyone with a history of substance abuse.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Change in Skin and Hair Health Assessed by Dermatologist Evaluation | Baseline to Week 12
  Assessment of changes in skin and hair health from baseline to Week 12 based on standardized digital photographs evaluated by a dermatologist.

SECONDARY OUTCOMES:
Change in Participant-Reported Nail Strength, Joint Mobility, and Well-Being | Baseline, Week 2, Week 4, Week 8, and Week 12
  Self-reported changes in nail strength, joint health, muscle recovery, and overall well-being measured via study-specific online questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States